CLINICAL TRIAL: NCT03098498
Title: Impact of Debridement Invasiveness on Attachment Gain After Antiinfective Periodontal Therapy
Acronym: ATTGAIN16
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ulrich Schlagenhauf, Chairman Dept. of Periodontology, Wuerzburg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WuerzburgUH
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Periodontitis; Periodontal Attachment Loss; Periodontal; Lesion
Keywords: periodontitis; scaling; attachment gain; air polishing; periodontal lesion
MeSH Terms: conditions — Periodontitis; Periodontal Attachment Loss | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: controlled prospective parallel group intervention trial
Who Masked: Outcomes Assessor
Masking Description: The examiner performing the assessment of periodontal attachment gain is not aware of the type of the preceding intervention therapy (one-stage vs. two-stage) provided to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two-Stage Subgingival Debridement (Experimental): Initially soft subgingival bacterial biofilms are removed from periodontal lesions by an airpolishing device and erythritol cleaning powder. 6 weeks later subgingival calculus is mechanically removed in a second step by mechanical scaling and root planing
  Interventions: Procedure: Subgingival Debridement
- One-Stage Subgingival Debridement (Active Comparator): Soft subgingival bacterial biofilms, as well as subgingival calculus are concomitantly removed from periodontal lesions by mechanical scaling and root planing
  Interventions: Procedure: Subgingival Debridement

INTERVENTIONS:
Procedure: Subgingival Debridement — Removal of subgingival bacterial biofilms and subgingival calculus from periodontal lesions
  Other Names: Scaling and Root Planing

SUMMARY:
This study compared the gain of periodontal attachment after concomitant one-stage removal of bacterial biofilms and subgingival calculus with a two-stage procedure removing subgingival calculus 6 weeks after the initial removal of soft subgingival bacterial biofilms.

DETAILED DESCRIPTION:
The concomitant removal of subgingival calculus and soft bacterial biofilms in a one-stage procedure might impair periodontal healing in deep infrabony pockets due to the mechanical disruption of demineralized bone sections at the bottom of periodontal lesions. This randomized controlled clinical trial therefore aims at comparing the resulting attachment gain 6 months after one-stage antiinfective periodontal therapy comprising the concomitant subgingival removal of soft bacterial biofilms and calculus with a two-stage approach removing subgingival calculus only 6 weeks after the initial removal of soft subgingival bacterial biofilms.

ELIGIBILITY:
Inclusion Criteria:

* presence of periodontal disease
* minimum of 1 tooth with an infrabony periodontal lesion and pocket depth ≥ 6mm
* minimum of 15 natural teeth

Exclusion Criteria:

* systemic disease interfering with periodontal healing (e.g. diabetes)
* antibiotic therapy ≤ 12 month prior to study participation
* necessity for preventive antibiotic therapy during dental interventions
* inability to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schlagenhauf, Prof. Dr., Principal Investigator — Chairman Dept. of Periodontology, University Hospital Wuerzburg, Germany
Locations (1):
- Dept. of Periodontology, University Hospital Wuerzburg, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Two-Stage Subgingival Debridement | One-Stage Subgingival Debridement
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Two-Stage Subgingival Debridement | One-Stage Subgingival Debridement | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 63.5 (6.8) | 58.4 (9.2) | 61.0 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 22 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Attachment Loss
Description: Difference in millimeter (mm) in the distance between the cemento-enamel-junction and the probable bottom of the periodontal pocket recorded at baseline and at the end of the study in periodontal pockets with a baseline pocket depth ≥ 6 mm
Time Frame: 168 days (24 weeks)
Population: patients suffering from untreated severe chronic periodontitis
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Two-Stage Subgingival Debridement | One-Stage Subgingival Debridement
Number analyzed (Participants) | 22 | 22
mm | -1.08 (1.26) | -1.22 (0.90)

2. Secondary Outcome: Change in Bleeding on Probing
Description: Difference in the mean percentage of probed periodontal probing sites in teeth with initial pocket depth ≥ 6 mm displaying bleeding on probing between baseline and end of the study.
Time Frame: 168 days (24 weeks)
Population: patients suffering from untreated severe chronic periodontitis
Measure: Mean (Standard Deviation); unit: percentage of bleeding sites
Arm/Group | Two-Stage Subgingival Debridement | One-Stage Subgingival Debridement
Number analyzed (Participants) | 22 | 22
percentage of bleeding sites | -10 (40) | -20 (41)

3. Secondary Outcome: Change in Probing Pocket Depth
Description: Difference in probing pocket depth between baseline and end of study in teeth with a baseline periodontal probing pocket depth ≥ 6 mm
Time Frame: 168 days (24 weeks)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Two-Stage Subgingival Debridement | One-Stage Subgingival Debridement
Number analyzed (Participants) | 22 | 22
mm | -1.53 (0.99) | -1.17 (0.92)

4. Secondary Outcome: Change in Gingival Index (GI)
Description: Measuring the mean difference in Gingival Index (GI) scores between baseline and end of the study
Time Frame: 168 days (24 weeks)
Population: In deviation from the original study protocol, the GI values were not recorded, as bleeding on probing is the relevant measure for assessing the extent of gingival inflammation according to the current classification adopted by the EFP/AAP.
Arm/Group | Two-Stage Subgingival Debridement | One-Stage Subgingival Debridement
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Plaque Index
Description: Measuring the difference in the extent of supragingival plaque coverage according to the criteria set by Silness and Loe between baseline and end of study
Time Frame: 168 days (24 weeks)
Measure: Mean (Standard Deviation); unit: % of tooth surfaces
Arm/Group | Two-Stage Subgingival Debridement | One-Stage Subgingival Debridement
Number analyzed (Participants) | 22 | 22
% of tooth surfaces | -18 (30) | -8 (34)

ADVERSE EVENTS:
Time Frame: Occurring adverse event data were collected from baseline to the end of study (168 days).
Arm/Group | Two-Stage Subgingival Debridement | One-Stage Subgingival Debridement
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT03098498/Prot_SAP_000.pdf